CLINICAL TRIAL: NCT05511454
Title: Comparison of Salivary and Crevicular Protein Concentrations of FIBA, PLMN, HEMO and ApoH in Healthy and Periodontitis Patients
Acronym: PerioBioTIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0067
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Periodontitis; Periodontal Diseases
Keywords: Periodontitis; Proteome; ELISA test; Biomarkers
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Pilot pathophysiological study of comparative ELISA proteomic analysis of salivary and crevicular samples in periodontitis patients vs. control subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of patients with periodontitis (cases) (Experimental): Patients with periodontitis according to the Chicago 2018 classification criteria
  Interventions: Other: Salivary and crevicular samples
- Control group (Other): Patients with periodontal health according to the 2018 Chicago Classification
  Interventions: Other: Salivary and crevicular samples

INTERVENTIONS:
Other: Salivary and crevicular samples — The samples will be taken from patients in both groups who meet the selection criteria during consultations at the Montpellier University Hospital's Odontology Department. During these consultations, a sample will be taken after rinsing the oral cavity with a glass of water. The samples will be taken before the periodontal assessment in order to avoid bleeding.

SUMMARY:
Periodontal disease is a multifactorial inflammatory disease of infectious origin. The last epidemiological study concerning periodontitis in France was carried out in 2002-2003 by Bourgeois et al and shows that 95.4% of the patients have a loss of attachment and 82.23% have associated periodontal pockets. The presence of bacteria, mostly Gram-negative anaerobes, is not sufficient to explain the heterogeneity of clinical forms. Indeed, there are different risk factors influencing the frequency and severity of periodontitis.

Moreover, the link between systemic pathologies and periodontitis has been widely established: it concerns metabolic syndromes, cardiovascular pathologies, premature pregnancies, autoimmune diseases and Alzheimer disease.

Some research has been done on biomarkers found in periodontitis. Among them, the investigators quote the study which took place within the laboratory of Biochemistry - Clinical Proteomics of Pr Lehmann Sylvain by Mertens et al. It is the only study to date that has established an LC-MRM proteomic profile characteristic of periodontitis: indeed, 4 proteins of plasma origin were highlighted thanks to this technology: hemopexin (HEMO), plasminogen (PLMN), apolipoprotein H and α-fibrinogen (FIBA) were correlated with the presence of periodontitis compared to the control group (p<0.05).

DETAILED DESCRIPTION:
Periodontitis can be defined as a multi-factorial infectious disease, initiated by the accumulation of bacterial biofilm on the dental surfaces and causing the destruction of the supporting tissues of the tooth, which can lead to the loss of the dental organ. The high prevalence of these pathologies in the general population makes them an important subject to be considered in public health. This prevalence varies from 56 to 82%. The last epidemiological study in France carried out in 2002-2003 shows that 95.4% of patients have a loss of attachment and 82.23% have associated periodontal pockets. They are related to an imbalance between the microbiota and the host which will be more or less permissive with respect to the quantity and/or the bacterial quality. The presence of bacteria, mostly Gram-negative anaerobes, is not sufficient to explain the heterogeneity of clinical forms. Indeed, undetermined etiological factors create in some patients an environment favorable to the formation of periodontitis, in particular genetic and predisposing factors.

Periodontitis is characterized by variable clinical symptoms and signs that may include visible or non-visible inflammation, spontaneous or provoked gingival bleeding of varying severity, periodontal pocket formation related to attachment and alveolar bone loss, tooth mobility and may lead to tooth loss. In practice, the diagnosis is based on the new Chicago classification but the etiological diagnosis is not so simple with the clinical and radiological tools available today. Bacteriological tests exist to identify certain bacteria responsible for periodontitis, but here again these tests are not sufficiently effective and studies show that there is a significant risk of false positives and negatives.

Some research has been done on biomarkers found in periodontitis. The PubMed database includes a few articles on salivary biomarkers and periodontitis, including a systematic review dating from 2018. Among them, the investigators mention the study that took place in the laboratory of Biochemistry - Clinical Proteomics of Pr Lehmann Sylvain by Mertens et al. It is the only study to date that has established an LC-MRM proteomic profile characteristic of periodontitis: indeed 4 proteins of plasma origin were highlighted thanks to this technology: hemopexin (HEMO), plasminogen (PLMN), apolipoprotein H and α-fibrinogen (FIBA) were correlated to the presence of periodontitis compared to the control group (p<0.05).

* PLMN: lower level in periodontitis patients than in control patients.
* HEMO and FIBA: higher levels in samples from patients with aggressive periodontitis.
* Apolipoprotein H has been identified as a differential diagnosis between aggressive and chronic periodontitis. Its level is significantly higher in patients with aggressive periodontitis.
* All proteins correlated with periodontal disease are proteins of plasma origin

However, this study is only interested in saliva. However, the proteins found are of plasma origin. The crevicular fluid (present in the sulcus) is a plasma exudate that is easy to collect. More and more studies are interested in this fluid. It would therefore be interesting to analyze it in parallel with saliva.

This assay of proteins in fluids can detect a maximum of 4 to 5 proteins in a multiplex assay, and requires prior knowledge of the proteins being sought. In order to open up the search for new biomarkers, quantification techniques using mass spectrometry coupled with high-performance liquid chromatography provide extensive qualitative and quantitative characterisation of the peptidome and epitranscriptome. Nowadays, with the DIA (Data Independent Acquisition) mode, multiplex detection can be extended to more than 1000 proteins in a single analysis, as shown in a recent study by Sato et al. The advantages of these techniques lie in their high specificity and sensitivity, enabling the detection of thousands of proteins and multiple RNA modifications in micro-samples (microlites).

ELIGIBILITY:
Inclusion Criteria:

Control Group:

* Patients consulting the Center for Dental Care, Education and Research for the care of their periodontal pathology.
* Patients with periodontal health according to the 2018 Chicago Classification.

Case Group:

* Patients consulting the Center for Dental Care, Education and Research for the care of their periodontal pathology.
* Patients with periodontitis according to the Chicago 2018 classification criteria.

Exclusion Criteria:

General:

* Pregnancy in progress or planned during the study period, Pregnant or breastfeeding women.
* Adult protected by law or patient under tutorship or curatorship.
* Participation in other ongoing biomedical research.
* Failure to obtain written informed consent after a reflection period.
* Not be affiliated to a French social security system or a beneficiary of such a system.

Case Group:

* Patients with previous periodontal treatment or maintenance.

Control Group:

* There is no prohibition against subjects participating in other research simultaneously.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-12-22 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of plasma protein concentration between the two groups | 1 day
  Salivary and crevicular concentrations of each of the plasma proteins (FIBA, PLMN, ApoH, HEMO), measured by ELISA in the case and control groups (in µg/mL). Salivary and crevicular samples will be analyzed using specific ultra-sensitive Meso Scale Discovery (MSD) immunoassay kits.

SECONDARY OUTCOMES:
Comparison of plasma protein concentration according to the stages and grades of periodontitis (in case group). | 1 day
  Salivary and crevicular concentrations of each of the plasma proteins (FIBA, PLMN, ApoH, HEMO), measured by ELISA in the case group according to the stages and grades of periodontitis stated by the Chicago 2018 classification (in µg/mL). Salivary and crevicular samples will be analyzed using specific ultra-sensitive Meso Scale Discovery (MSD) immunoassay kits.
Comparison of plasma protein concentration according to the presence or absence of diabetes (in case group). | 1 day
  Salivary and crevicular concentrations of each of the plasma proteins (FIBA, PLMN, ApoH, HEMO), measured by ELISA in the case group according to the presence or absence of diabetes (in µg/mL). Salivary and crevicular samples will be analyzed using specific ultra-sensitive Meso Scale Discovery (MSD) immunoassay kits.
Quantitative measure | 1 day
  Concentrations of each of the plasma proteins (FIBA, PLMN, ApoH, HEMO), measured by ELISA in salivary samples and in crevicular samples (in µg/mL). Salivary and crevicular samples will be analyzed using specific ultra-sensitive Meso Scale Discovery (MSD) immunoassay kits.
Comparison of salivary and crevicular protein profiles and protein levels after mass spectrometry analysis between subjects with periodontitis and a control group | 1 day
  Salivary and crevicular concentrations of each of the plasma proteins (FIBA, PLMN, ApoH, HEMO), measured by mass spectrometry analysis for subjects with periodontitis and a control group.
Comparison of level of free nucleosides found in saliva and crevicular fluid by mass spectrometry between subjects with periodontitis and a control group. | 1 day
  Comparison of salivary and crevicular epitranscriptomic profiles and free nucleoside levels after mass spectrometry analysis between subjects with periodontitis and a control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Soins Dentaires, Montpellier, France